CLINICAL TRIAL: NCT01025804
Title: Post-marketing Surveillance Study of the Pharmacokinetics of Asparaginase and Antibody Formation in Interfant-06
Brief Title: Pharmacokinetics of Asparaginase and Antibody Formation in Interfant-06
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Birgitte Klug Albertsen, MD, PhD, Aarhus University Hospital
Other Study IDs: Interfant-06, NOPHO; register identifier (Registry Identifier: NOPHO)
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Leukemia
Keywords: Interfant-06; Infant ALL; Asparaginase; Pharmacokinetics of asparaginase; Antibody formation
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum is retained for measurement of enzyme activities and antibodies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants

SUMMARY:
Asparaginase is an important drug in the treatment of childhood leukemia including in infant (<1 year). The prognosis for infants is bad.

Information about drug metabolism in neonates and infants is scarce as well as the reactions of an immature immune system to foreign proteins. The aims of this study is to describe the metabolism (pharmacokinetics) of asparaginase after administration intramuscularly and to evaluate the formation of antibodies against the drug (enzyme) during treatment in order to optimize the asparaginase treatment in infants in the future.

DETAILED DESCRIPTION:
Combination chemotherapy for acute lymphoblastic leukaemia (ALL) usually includes a bacterial L-asparaginase enzyme derived from Escherichia coli or Erwinia species. Several studies have described the pharmacokinetics in children above 1 year of age of asparaginase given intramuscularly as well as intravenously. The development of anti-asparaginase antibodies to these foreign proteins has also been described.

Chemotherapy for infant ALL also includes L-asparaginase. However, the pharmacokinetics of asparaginase and antibody formation in infants is needed to be described to optimize therapy for this group of patients who have a doubtful prognosis.

Background In general the information about drug metabolism in neonates and infants is scarce as well as the reactions of an immature immune system to foreign proteins. Several pharmacokinetic studies have been performed in children above one year of age, but no data is available about pharmacokinetics and antibody formation during treatment with any asparaginase preparation in infants.

Pharmacokinetics:

Asparaginase is used in the treatment of childhood ALL since it depletes the blood of asparagines, which can be synthesized by normal cells but not by leukemic lymphoblasts. It has been shown that serum activities above 100 IU/l ensure depletion of asparagine in serum and CNS. In many cases even values considerably lower than 100 IU/l will deplete asparagine from the serum1-5.

In the Interfant-06 protocol the doses of asparaginase are adopted from childhood ALL-protocols without scientific foundation. Infants may metabolise asparaginase differently and thus may not achieve amino acid depletion.

Antibody formation:

Asparaginase is a foreign protein for the human body, so patients may develop antibodies against it, resulting in allergic reactions (probably mediated by IgE-antibodies) or silent antibodies (IgG antibodies, blocking the effect of the enzyme). In the first case treatment most often is stopped and in the second case treatment is insufficient6-7, and thus giving the patient a poorer prognosis in both cases.

In Interfant-06 patients are treated with native E.coli asparaginase for a period followed by PEG-asparaginase later during their treatment. Studies in older children have shown that approximately 1/3 of the patients develop IgG-antibodies against native E.coli after 5-6 doses7. Other studies have shown that IgG-antibodies against native E.coli asparaginase cross-react with PEG-asparaginase, resulting in a faster clearance of the enzyme8. Allergic reactions (any grade) to native E.coli asparaginase are encountered in approximately 30 % of children11-12. There is no knowledge about the frequency of antibody formation during asparaginase therapy in infants.

Aim

The study has the purposes:

* to describe the pharmacokinetics of intramuscular native E.coli and PEG-asparaginase in children below 1 year at diagnosis
* to evaluate antibody formation during asparaginase treatment with E.coli followed by PEG-asparaginase in infants

ELIGIBILITY:
Inclusion Criteria:

* infants <1 year at diagnosis
* diagnosed with ALL
* treated according to the international Interfant-06 protocol
* treated at one of the pediatric oncological centers in the Nordic countries

Exclusion Criteria:

* children >1 year at diagnosis

Ages: 1 Hour to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants (children < 1 year) with ALL treated according to Interfant-06 at one of the Pediatric Oncology Centers in the Nordic Countries
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2009-12; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics, antibody formation, side effects | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte K Albertsen, MD, Study Chair
Locations (6):
- Denmark (2):
  - Aarhus University Hospital, Department of Pediatrics Skejby Hospital, Aarhus, Aarhus N
  - Rigshospitalet, Copenhagen
- Helsinki University Hospital, Helsinki, Finland
- University Hospital Reykjavik, Reykjavik, Iceland
- Rikshospitalet, Oslo, Norway
- Karolinska, Stockholm, Sweden

REFERENCES:
- [Derived] Albertsen BK, Harila-Saari A, Jahnukainen K, Lahteenmaki P, Riikonen P, Mottonen M, Lausen B. Asparaginase treatment in infants with acute lymphoblastic leukemia; pharmacokinetics and asparaginase hypersensitivity in Interfant-06. Leuk Lymphoma. 2019 Jun;60(6):1469-1475. doi: 10.1080/10428194.2018.1538507. Epub 2019 Jan 11. PMID 30632847